CLINICAL TRIAL: NCT00208442
Title: A Prospective, Randomised, Controlled, Single Centre, Blinded Study of the Wear Characteristics of Two Polyethylene Bearing Surfaces, Enduron vs. Marathon
Brief Title: A Randomised Single Centre Study to Compare the Long-term Wear Characteristics of Marathon™ and Enduron™ Polyethylene Cup Liners in Primary Total Hip Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT99/31
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis; Collagen Disorders; Avascular Necrosis; Traumatic Femoral Fractures; Nonunion of Femoral Fractures; Congenital Hip Dysplasia; Slipped Capital Femoral Epiphysis
Keywords: Hip; Cemented
MeSH Terms: conditions — Osteoarthritis; Collagen Diseases; Osteonecrosis; Hip Dislocation, Congenital; Slipped Capital Femoral Epiphyses

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marathon™ (Active Comparator): Moderately cross-linked polyethylene liner in a modular acetabular component
  Interventions: Device: Marathon™
- Enduron™ (Active Comparator): Standard UHMWPE polyethylene liner in a modular acetabular component
  Interventions: Device: Enduron

INTERVENTIONS:
Device: Marathon™ — Moderately cross-linked polyethylene liner in a modular acetabular component
  Arms: Marathon™
Device: Enduron — Standard polyethylene liner in a modular acetabular component
  Arms: Enduron™

SUMMARY:
The purpose of this study is to compare the performance and compare the wear characteristics of two polyethylene cup liners, Marathon™ and Enduron™, in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be randomly allocated to one of the polyethylene cup liners, Marathon™ or Enduron™ and will be evaluated at regular intervals using clinical and x-ray assessments.

DETAILED DESCRIPTION:
The original protocol intended to perform clinical assessment using the Harris Hip Score, Merle D'Aubigne score and UCLA Activity Level Rating at 6 months, 1 year, 2 years, 3 years, 4 years, 5 years and 10 years post-operative. Merle D'Aubigne score evaluation was removed per Amendment 2.

However, protocol-specified data collected included only the linear and volumetric wear and incidence and pattern of radiological signs at 10 years post surgery. Data collected outside of the protocol included Oxford Hip Score and SF-12 for mental and physical well-being at 10 years post surgery and revision for any reason.

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 45 and 75 years inclusive.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who, in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects with non-inflammatory arthritis of the hip who require a primary hip arthroplasty and are considered by the Clinical Investigator to be suitable for a cemented femoral component and an uncemented acetabular component.

v) Subjects who have a Charnley C classification

vi) Subjects who have undergone a contralateral hip replacement within past 6 months

vii) Subjects with a poorly functioning contralateral hip replacement or one which has been identified as requiring revision

viii) The first hip replacement scheduled for subjects identified as requiring primary bi-lateral hip replacements which will not be conducted simultaneously (i.e. on the same day).

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study.

ii) Women who are pregnant.

iii) Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.

iv) Subjects who have participated in a clinical study with an investigational product in the last month.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2001-06-01 (Actual); Primary Completion 2006-09-01 (Actual); Study Completion 2013-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the linear and volumetric wear at the three-year time point. | 10yrs post surgery

SECONDARY OUTCOMES:
Demonstrate the difference in the 3D femoral head displacement between Enduron™ and Marathon™ three-years post-operatively | 10yrs post surgery
Radiographic analysis | 10yrs post surgery
Oxford Hip Score | 10yrs post surgery
SF-12 for Mental and Physical well-being | 10yrs post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University Otago, Wellington Medical School of Medicine, Wellington, New Zealand

REFERENCES:
- [Result] Calvert GT, Devane PA, Fielden J, Adams K, Horne JG. A double-blind, prospective, randomized controlled trial comparing highly cross-linked and conventional polyethylene in primary total hip arthroplasty. J Arthroplasty. 2009 Jun;24(4):505-10. doi: 10.1016/j.arth.2008.02.011. Epub 2008 Jun 10. PMID 18547784
- [Result] Mutimer J, Devane PA, Adams K, Horne JG. Highly crosslinked polyethylene reduces wear in total hip arthroplasty at 5 years. Clin Orthop Relat Res. 2010 Dec;468(12):3228-33. doi: 10.1007/s11999-010-1379-4. PMID 20458640